CLINICAL TRIAL: NCT06151366
Title: Early Detection of Pulmonary Exacerbations in Non-cystic Fibrosis Bronchiectasis
Acronym: Bronch-EX
Status: Not yet recruiting | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: LifeArc (Other)
Responsible Party: Sponsor
Other Study IDs: P03012; 323297 (Other: IRAS)
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Non-cystic Fibrosis Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non interventional — non interventional

SUMMARY:
The goal of this observational study is to learn about the use of equipment to monitor health at home in participants who have non-cystic fibrosis bronchiectasis. The main question[s] it aims to answer are:

* How acceptable participants find using home monitoring equipment.
* To find out if the data collected from home monitoring can help to detect chest infections (exacerbations) before participants get symptoms they are aware of.

Participants will be provided with -

* a handheld spirometer to record FEV1 (lung function)
* a Fitbit, or other compatible activity monitor, to record activity and heart rate
* a saturation monitor that fits painlessly on the end of the finger to record oxygen levels
* weighing scales to record weight
* a mini freezer and pre-labelled sample containers to store a daily sputum sample. There is enough room in the freezers for samples to be brought to routine clinic visits. We will provide a cool bag and freezer packs for this. A courier collection of the samples can be arranged if necessary.

Participants will be encouraged to perform lung function, activity and oxygen levels at least 4 x per week.

Participants will be guided through how to set up and use each piece of equipment by the research team. The devices all connect to a smartphone app called Breathe RM (Remote Monitor,) which is free to download, via Bluetooth. Once set up using the home monitoring devices and adding notes to the app should take no more than 15 minutes per day.

Participants will be asked to record in the app -

* episodes of pulmonary exacerbation that require antibiotic treatment
* their coughing and wellness scores daily

DETAILED DESCRIPTION:
The aim of the study is to find out if data collected from home monitoring and artificial intelligence (AI) in patients with non-Cystic Fibrosis bronchiectasis can be used to detect pulmonary exacerbations (chest infections) before participants get symptoms of an infection. The infection can then be treated sooner and therefore potentially reduce long term lung damage. This study builds on previous work that has been done with patients who have a lung condition called cystic fibrosis and has shown favourable results. The AI technology relates to the predictive algorithm and not to any devices.

Potential participants will be approached during routine clinic visits (face to face or virtual) to offer more information regarding the study, provided with written and verbal information, given the opportunity to ask questions and given ample time to make a decision regarding whether or not they would like to take part.

Fifty patients from Royal Papworth Hospital who have a diagnosis of non-Cystic Fibrosis Bronchiectasis and who have a history of one or more pulmonary exacerbations in the previous year will be asked to perform home monitoring, record episodes of infection and provide a daily sputum sample for 6 months.

Participants will be provided with -

* a handheld spirometer to record Forced expiratory volume in 1 second (FEV1) (lung function)
* a Fitbit, or other compatible activity monitor, to record activity and heart rate
* a saturation monitor that fits painlessly on the end of the finger to record oxygen levels
* weighing scales to record weight
* a mini freezer and pre-labelled sample containers to store a daily sputum sample. There is enough room in the freezers for samples to be brought to routine clinic visits. We will provide a cool bag and freezer packs for this. A courier collection of the samples can be arranged if necessary.

Participants will be encouraged to perform lung function, activity and oxygen levels at least 4 x per week.

Participants will be guided through how to set up and use each piece of equipment by the research team. The devices all connect to a smartphone app called Breathe RM (Remote Monitor) (free to download) via Bluetooth. Once set up using the home monitoring devices and adding notes to the app should take no more than 15 minutes per day.

Participants will be asked to record in the app -

* episodes of pulmonary exacerbation that require antibiotic treatment
* coughing and wellness scores daily

We want to find out how participants find performing home monitoring and what impact it has on quality of life. To assess this we will ask participants to complete a questionnaire to find out how acceptable they find using the equipment and app at home and a questionnaire that gives information regarding quality of life. These questionnaires can be provided on paper or electronically depending on participant preference. They should take no more than 15 minutes each to complete. The acceptability questionnaire will be taken 3 months into the study and at the end of the study. The quality-of-life questionnaire will be taken at the start, middle and end of the study. If a participant withdraws they will be asked to perform the questionnaires at this time.

Participants who use a nebuliser will be given the option to change to a Pari eFlow rapid nebuliser with Pari Connect. The nebuliser connects to an app on their smartphone via Bluetooth and monitors how often the participant takes their inhaled medications. Participants will be guided through how to use this equipment.

A score of how breathless participants (MRC Dyspnoea Scale) are and how severe the bronchiectasis (Bronchiectasis Severity Index) is will be performed at the start and end of the study by the clinical or research team and takes a few minutes.

Participants will be invited to virtual groups or one to one discussions to give feedback to the research team regarding the experience of being on the study. This is voluntary and participants will not be identified when the study is written up for publication.

Participants will be provided with a phone number and email address to contact the research team during office hours with any study related issues. All clinical queries should be directed to the clinical team as usual. Participants can withdraw at any time and it will have no impact on their care.

Results of the study will be made available through email, text, newsletters, hospital social media and virtual group / individual discussions.

ELIGIBILITY:
Inclusion Criteria:

* Under the care of the Lung Defence Clinic at Royal Papworth Hospital
* CT confirmed diagnosis of bronchiectasis
* Age >/= 18 years
* Had two or more clinician defined APEs in the year prior to enrolment
* Typically expectorates sputum daily
* Considered suitable for home monitoring in the opinion of the investigator
* Able to provide written informed consent

Exclusion Criteria:

* Patients unable to provide written informed consent
* Known cystic fibrosis
* Lung transplant recipients or on lung transplant waiting list
* Use of long-term oxygen therapy (LTOT) or non-invasive ventilation to manage respiratory failure
* Patients unwilling to consent to their link anonymised data from home monitoring being used for research
* Patients unable to use a smartphone. Patients who would like to take part but do not have a smartphone can be provided with one.
* Patients who do not have reliable Wi-Fi at home or are unable to access public Wi-Fi at least twice per week.
* Considered unsuitable for home monitoring in the opinion of the investigator

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Under the care of the Lung Defence Clinic at Royal Papworth Hospital
  * CT confirmed diagnosis of bronchiectasis
  * Age >/= 18 years
  * Had two or more clinician defined APEs in the year prior to enrolment
  * Typically expectorates sputum daily
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in the bronchiectasis impact measure scores at 6 months compared to baseline | baseline and month 6
  The Bronchiectasis Impact Measure is a validated, patient reported outcome measure across 8 domains (cough, sputum, breathlessness, tiredness, activity, general health, control, exacerbations) and the impact they have on daily life. It is measured on a scale on 0 to 10 with 0 being no impact on daily life and 10 being greatly impacts daily life (lower score better). Minimum score 0 maximum score 10. Higher score mean worse outcome.

SECONDARY OUTCOMES:
The acceptability of home monitoring in participants with non-cystic fibrosis bronchiectasis | 3 months and 6 months
  Comparison of user acceptance questionnaire scores at 3 and 6 months. This is on a 5 point Likert scale with 5 being least acceptable and 1 being most acceptable. Higher score means worse outcomes.
Impact of home monitoring on acute exacerbation frequency | In preceding 12 months and at 6 months
  Number of days requiring antibiotics for acute pulmonary exacerbation at baseline and 6 months. Minimum score 0. Maximum score 365. Higher score means worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Papworth Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The current data sharing plans for this study are unknown and will be available at a later date